CLINICAL TRIAL: NCT00941993
Title: First in Man Evaluation of the Anesthetic Effect of Lidocaine/Epinephrine Solution Delivered Via Iontophoresis to the External Auditory Apparatus (FIM Iontophoresis Study)
Brief Title: Anesthetic Effect of Lidocaine/Epinephrine Solution Delivered Via Iontophoresis to External Auditory Apparatus
Acronym: IONTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPR005000
Record Dates: First submitted 2009-07-14; First posted 2009-07-20 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Acute Otitis Media; Chronic Otitis Media; Recurrent Acute Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- local anesthesia (Experimental): tympanic membrane local anesthesia delivery system
  Interventions: Device: Iontophoresis System (Acclarent)

INTERVENTIONS:
Device: Iontophoresis System (Acclarent) — Iontophoresis system will deliver iontophoresis simultaneously to both ears. Active elements of this drug delivery system are lidocaine and epinephrine.
  Other Names: Acclarent

SUMMARY:
This is a non-randomized, multicenter, prospective, clinical study intended to evaluate the effectiveness of a method for iontophoretic delivery of a buffered lidocaine/epinephrine solution for provision of tympanic membrane anesthesia in patients who are indicated for an ear procedure requiring penetration of the tympanic membrane, including, but not limited to, myringotomy, tympanocentesis with culture or tympanostomy with tube placement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 months and older
2. Both male and female patients eligible
3. Patients are indicated for procedures requiring penetration of the tympanic membrane (including, but not limited to, myringotomy, tympanocentesis with culture or tympanostomy with tube implant)

Exclusion Criteria:

1. Patients with a history of sensitivity or reaction to lidocaine, epinephrine or any hypersensitivity to local anesthetics of the amide type or any component of the drug solution
2. Markedly atrophic, retracted, atelectatic or perforated tympanic membrane
3. Otitis externa
4. Electrically sensitive patients and patients with electrically sensitive support systems (pacemakers, defibrillators, etc.)
5. Damaged or denuded skin in the auditory canal
6. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry "Fritz" Butehorn, III, MD, Principal Investigator — Spartanburg ENT
Locations (1):
- Spartanburg ENT, Spartanburg, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Iontophoretic Delivery of Local Anesthesia: Tympanic membrane anesthesia delivery system
  Iontophoresis System (Acclarent) : Iontophoresis system will deliver iontophoresis simultaneously to both ears. Active elements of this drug delivery system are lidocaine and epinephrine.
Period: Overall Study
Arm/Group | Iontophoretic Delivery of Local Anesthesia
Started | 109
Completed | 109
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Iontophoretic Delivery of Anesthesia: Tympanic membrane anesthesia delivery system
  Iontophoresis System (Acclarent) : Iontophoresis system will deliver iontophoresis simultaneously to both ears. Active elements of this drug delivery system are lidocaine and epinephrine.
Arm/Group | Iontophoretic Delivery of Anesthesia
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.0 (22.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieved Anesthesia Effectiveness Per Investigator Assessment
Description: Investigator performed a gentle tap of the tympanic membrane to assess whether adequate anesthesia was achieved following local anesthesia by iontophoresis. All subjects for which an ear procedure was attempted were considered to have achieved anesthesia effectiveness.
Time Frame: Day 0
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Anesthesia: tympanic membrane anesthesia delivery system
  Iontophoresis System (Acclarent) : Iontophoresis system will deliver iontophoresis simultaneously to both ears. Active elements of this drug delivery system are lidocaine and epinephrine.
Arm/Group | Anesthesia
Number analyzed (Participants) | 109
percentage of subjects | 89.9 [82.7 to 94.9]

2. Secondary Outcome: Patient Tolerability of Iontophoresis Procedure Will be Measured Using a Wong Baker Faces Pain Scale
Description: Includes all subjects for whom Iontophoresis current delivery was initiated.
  The Wong-Baker FACES pain scoring system is a scale of 0 to 5, where 0 means 'no hurt', 1 = 'hurts a little bit', 2 = 'hurts little more', 3 = 'hurts even more', 4 = 'hurts whole lot' and 5 = 'hurts worst'.
  The Wong-Baker scores are reported by subject.
Time Frame: Day 0
Population: Analysis population includes subjects completing iontophoresis for which Wong Baker scores are available.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Anesthesia: tympanic membrane anesthesia delivery system
  Iontophoresis System (Acclarent): Iontophoresis system will deliver iontophoresis simultaneously to both ears. Active elements of this drug delivery system are lidocaine and epinephrine.
Arm/Group | Anesthesia
Number analyzed (Participants) | 101
units on a scale | 0.7 (1.2)

3. Secondary Outcome: Subject/Parent Reported Satisfaction With the In-office Procedure
Description: Adult subjects or parents of pediatric subjects were asked to rate their agreement or disagreement with the statement: 'Overall, I am satisfied with the whole procedure'. Response options included: 'Strongly Disagree', 'Disagree', 'Neutral', 'Agree' or 'Strongly Agree'. The number of respondents who reported that they 'agree' or 'strongly agree' that they were satisfied with the whole procedure are reported.
  The analysis population does not include the full study cohort as this survey question was implemented during, not prior to, the enrollment period.
Time Frame: Day 0
Measure: Number (95% Confidence Interval); unit: % adult subjects or parents
Arm/Group | Anesthesia
Number analyzed (Participants) | 87
% adult subjects or parents | 94.3 [87.1 to 98.1]

4. Other Pre Specified Outcome: Patient Tolerability of In-office Ear Treatment Using the Wong Baker FACES Pain Scale.
Description: The Wong-Baker FACES pain scoring system is a subject-reported instrument using a scale of 0 to 5, where 0 means 'no hurt', 1 = 'hurts a little bit', 2 = 'hurts little more', 3 = 'hurts even more', 4 = 'hurts whole lot' and 5 = 'hurts worst'.
  Pain scores were recorded for all subjects for which an ear procedure was attempted.Pain scores are presented by subject, as an average of pain scores for both ears.
Time Frame: Day 0
Population: Analysis population includes subjects who completed anesthesia and for which an ear procedure was attempted
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anesthesia
Number analyzed (Participants) | 99
units on a scale | 1.0 (1.5)

5. Primary Outcome: Evaluate Any Adverse Effects Associated With the Iontophoresis System (Adverse Device Effects).
Time Frame: Day 0
Measure: Number; unit: participants
Arm/Group | Anesthesia
Number analyzed (Participants) | 109
participants
  Vertigo | 1
  Mild erythema at return electrode | 1

ADVERSE EVENTS:
Time Frame: 1 day (day of procedure)
Arm/Group | Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 2/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anesthesia (N=109)
Vertigo (Nervous system disorders) | 1 (1)
Mild Erythema at return electrode (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days